CLINICAL TRIAL: NCT03683030
Title: Safety and Effectiveness Evaluation of the Multi-Electrode Radiofrequency Balloon Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation (STELLAR)
Brief Title: Safety and Effectiveness Evaluation of the Multi-Electrode Radiofrequency Balloon Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation
Acronym: STELLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI_2017_04
Record Dates: First submitted 2018-09-14; First posted 2018-09-25 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
Keywords: Interventional; Radiofrequency Ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Group (Experimental): Ablation using Multi-electrode Radiofrequency (RF) Balloon Catheter (HELIOSTAR).
  Interventions: Device: Multi-Electrode RF Balloon Catheter

INTERVENTIONS:
Device: Multi-Electrode RF Balloon Catheter — Multi-Electrode RF Balloon Catheter will be inserted
  Other Names: HELIOSTAR

SUMMARY:
The primary objective of this clinical investigation is to demonstrate safety and effectiveness of the Multi-Electrode RF Balloon catheter for the treatment of drug refractory symptomatic paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The STELLAR study is a pivotal, prospective, multicenter, single-arm, clinical evaluation of the Multi-Electrode RF Balloon catheter. The study will evaluate the safety and effectiveness of the Multi-Electrode RF Balloon catheter used for ablation in patients with paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with Symptomatic Paroxysmal Atrial Fibrillation.

  1. At least two symptomatic AF episodes within last six months from enrollment.
  2. At least one ectrocardiographically documented AF episode within twelve (12) months prior to enrollment.
* Failed at least one Class I or Class III antiarrhythmic drug.
* Age 18 -75 years.

Key Exclusion Criteria:

* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
* Previous surgical or catheter ablation for AF.
* Previously diagnosed with persistent or long-standing persistent AF and/or Continuous AF > 7 days.
* Any percutaneous coronary intervention within the past 2 months.
* Valve repair or replacement or presence of a prosthetic valve.
* Any carotid stenting or endarterectomy within the past 6 months.
* Coronary artery bypass grafting, cardiac surgery, or valvular cardiac surgical procedure within the past 6 months.
* Documented left atrium (LA) thrombus within 1 day prior to the index procedure.
* LA antero posterior diameter > 50 mm.
* Left Ventricular Ejection Fraction (LVEF) < 40%.
* Contraindication to anticoagulation (e.g., heparin).
* Myocardial infarction within the past 2 months.
* Documented thromboembolic event (including transient ischemic attack) within the past 12 months.
* Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV.
* Awaiting cardiac transplantation or other cardiac surgery within the next 12 months.
* Presence of implanted pacemaker or implantable cardioverter defibrillator (ICD).
* Women who are pregnant, lactating, or who are of child bearing age and plan on becoming pregnant during the course of the clinical investigation.
* Life expectancy or other disease processes likely to limit survival to less than 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Srinivas Dukkipati, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Moussa Mansour, MD, Principal Investigator — Massachusetts General Hospital; J. Brian Deville, MD, Principal Investigator — Baylor Research Institute; Sandeep Goysl, MD, Principal Investigator — Piedmont Hospital; Arash Aryana, MD, Principal Investigator — Mercy General Hospital; Javier Roman-Gonzalez, MD, Principal Investigator — Methodist Texsan Hospital; Hugh Calkins, MD, Principal Investigator — Johns Hopkins University; Suneet Mittal, MD, Principal Investigator — The Valley Hospital; Bradley Knight, MD, Principal Investigator — Northwestern Memorial Hospital; Anshul Patel, MD, Principal Investigator — Emory St Joseph's Hospital; Sung Lee, MD, Principal Investigator — Medstar Health Research Institute; Douglas Packer, MD, Principal Investigator — Mayo Clinic; Michael Panutich, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian; Robert Sangrigoli, MD, Principal Investigator — Doylestown Hospital; Sharon Shen, MD, Principal Investigator — Vanderbilt Medical Center; Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Arrhythmia Research; Haseeb Jafri, MD, Principal Investigator — Kettering Medical Center; Timothy Mahoney, MD, Principal Investigator — Morristown Medical Center; Stavros Mountantonakis, MD, Principal Investigator — Lenox Hill Hospital; Massimo Grimaldi, MD, Principal Investigator — Miulli General Hospital; James Freeman, MD, Principal Investigator — Yale New Haven Hospital; Andy Voigt, MD, Principal Investigator — University of Pittsburgh Medical Center; Venkata Sagi, MD, Principal Investigator — Baptist Health Research Institute; Anil Bhandari, MD, Principal Investigator — University of Southern California; Haroon Rashid, MD, Principal Investigator — Inova Health Care Services; Naushad Shaik, MD, Principal Investigator — AdventHealth Orlando; Alan Wimmer, MD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri; Frank Cuoco, MD, Principal Investigator — Trident Medical Center; Madhu Reddy, MD, Principal Investigator — University of Kansas Medical Center; Ryan Aleong, MD, Principal Investigator — University of Colorado, Denver; Andre Gauri, MD, Principal Investigator — Spectrum Health System; Raul Weiss, MD, Principal Investigator — Ohio State University; Craig Cameron, MD, Principal Investigator — Oklahoma Heart; MArwan Bahu, MD, Principal Investigator — Phoenix Cardiovascular Research Group; Darryl Wells, MD, Principal Investigator — Swedish Medical Center; Ethan Ellis, MD, Principal Investigator — Med Center of the Rockies; Carlo Pappone, MD, Principal Investigator — Policlinico Di San Donato Milanese; Abdi Rasekh, MD, Principal Investigator — CHI Baylor St. Lukes Medical Center; Liqun Wu, MD, Principal Investigator — Ruijin Hospital; Chenyang Jiang, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (41):
- United States (37):
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Mercy General Hospital, Sacramento, California
  - University Of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Med Center of the Rockies, Loveland, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Health Research Institute, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory St Joseph's Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Arrhythmia Research, Overland Park, Kansas
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health System, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lenox Hill Hospital - Northwell Health, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Oklahoma Heart, Tulsa, Oklahoma
  - Doylestown Hospital, Doylestown, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - CHI Baylor St. Lukes Medical Center, Houston, Texas
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Inova Health Care Services, Falls Church, Virginia
  - Swedish Medical Center, Seattle, Washington
- China (2):
  - Ruijin Hospital, Rui Jin Er Road, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
- Italy (2):
  - Policlinico Di San Donato Milanese, Milanesi, MI
  - Ospedale "F. Miulli", Bari

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Goyal SK, Pappone C, Grimaldi M, Lee SW, Mountantonakis S, DeVille JB, Sagi VS, Jiang CY, Jafri H, Wimmer AP, Wu LQ, Dukkipati S, Rashid H, Calkins H, Mansour M, Roman-Gonzalez J, Natale A, Ciconte G, Aryana A; STELLAR investigators. Multielectrode Radiofrequency Balloon Catheter for Paroxysmal Atrial Fibrillation: Results From the Global, Multicenter, STELLAR Study. J Cardiovasc Electrophysiol. 2025 Feb;36(2):376-386. doi: 10.1111/jce.16524. Epub 2024 Dec 16. PMID 39686569

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per protocol, enrolled participants who had signed informed consent form but did not meet eligibility criteria prior to insertion of the study catheter were considered as screen failures and excluded from analysis.
Groups:
- Roll-in Phase: Participants enrolled in the roll-in phase with drug refractory, symptomatic paroxysmal atrial fibrillation (PAF) and were treated with the HELIOSTAR catheter in conjunction with the LassoStar catheter and Mutli-Channel radiofrequency (RF) Generator.
- Main Study: Participants enrolled in the main phase with drug refractory, symptomatic PAF, met eligibility criteria and had insertion of the HELIOSTAR catheter (with or without delivery of RF) in conjunction with the LassoStar catheter and Multi-Channel RF Generator.
Period: Overall Study
Arm/Group | Roll-in Phase | Main Study
Started (Enrolled participants) | 117 | 280
Evaluable Participants (Participants who were enrolled and had study catheter inserted) | 94 | 260
Completed | 93 | 249
Not Completed | 24 | 31
Not completed — Enrolled but screen failures | 12 | 7
Not completed — Enrolled but no catheter inserted | 11 | 13
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Early termination by subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 6
Not completed — Death | 0 | 2
Not completed — Catheter inserted but did not undergo ablation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Roll-in arm: Roll-in analysis set defined as all participants who were enrolled in the roll-in phase and had undergone the radiofrequency (RF) delivery with the study catheters. Main study arm: Modified intent-to-treat (mITT) analysis set defined as enrolled participants who met eligibility criteria and had insertion of the Biosense Webster HELIOSTAR catheter.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roll-in Phase | Main Study | Total
Number analyzed (Participants) | 94 | 257 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.30) | 60.1 (9.13) | 60.7 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 90 | 126
  Male | 58 | 167 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 36 | 40
  Not Hispanic or Latino | 78 | 193 | 271
  Unknown or Not Reported | 12 | 28 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 20 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 80 | 211 | 291
  Unknown or Not Reported | 7 | 19 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Primary Adverse Events (PAE) That Occurred Within 7 Days Following Atrial Fibrillation (AF) Ablation Procedure Using HELIOSTAR Catheter
Description: An AE is any untoward medical occurrence in a participant whether or not related to the investigational medical device. PAEs included myocardial infarction, thromboembolism, transient ischemic attack, phrenic nerve paralysis, major vascular access complication/bleeding, pericarditis, pulmonary edema (respiratory insufficiency), stroke/cerebrovascular accident (CVA), hospitalization (initial or prolonged), device or procedure related death, atrio-esophageal fistula, pulmonary vein stenosis.
Time Frame: Within 7 days post-procedure (Day of procedure = Day 0)
Population: Roll-in arm: Roll-in analysis set- participants who were enrolled in the roll-in phase and had undergone the radiofrequency (RF) delivery with the study catheters. Main study arm: Modified intent-to-treat (mITT) analysis set- enrolled participants who met eligibility criteria and had insertion of the Biosense Webster HELIOSTAR catheter. N (overall number of participants analyzed): participants evaluable for this outcome measure. Participants with missing values were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 94 | 255
Participants | 4 | 13

2. Primary Outcome: Number of Participants With Effectiveness Success
Description: Effectiveness success was defined as freedom from documented asymptomatic and symptomatic atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL; of unknown origin) episodes based on electrocardiographic data (greater than equal to [>=] 30 seconds on arrhythmia monitoring device) through the effectiveness evaluation period (Day 91 through Day 365 post index procedure) and freedom from the following failure modes : freedom from acute procedural failure, freedom from non-study catheter failure, freedom from repeat ablation failure, freedom from direct Current (DC) cardioversion failure, freedom from recurrence (captured on 12-lead electrocardiogram [ECG]) failure, and freedom from anti-arrhythmic drug failure. AFL of unknown origin was defined as all AFL except those Cavo-Tricuspid Isthmus (CTI) dependent AFL as confirmed by accepted electrophysiology (EP) maneuvers (example, entrainment or activation mapping) in an EP study.
Time Frame: From Day 91 up to Day 365 post-procedure (Day of procedure = Day 0)
Population: Roll-in arm: Roll-in analysis set defined as all participants who were enrolled in the roll-in phase and had undergone the RF delivery with the study catheters. Main study arm: mITT analysis set defined as enrolled participants who met eligibility criteria and had insertion of the Biosense Webster HELIOSTAR catheter. Here, N (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 94 | 250
Participants | 62 | 170

3. Secondary Outcome: Percentage of Participants With Acute Procedural Success
Description: Acute procedural success is defined as confirmation of entrance block in clinically relevant pulmonary veins (PVs) (all PVs except those that were silent and/or could not be cannulated) after adenosine and/or isoproterenol challenge (with or without the use of a focal catheter).
Time Frame: Day 0 (day of procedure)
Population: Roll-in arm: Roll-in analysis set defined as all participants who were enrolled in the roll-in phase and had undergone the RF delivery with the study catheters. Main study arm: mITT analysis set defined as enrolled participants who met eligibility criteria and had insertion of the Biosense Webster HELIOSTAR catheter. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 94 | 256
percentage of participants | 100 | 98.8

4. Secondary Outcome: Percentage of Participants With Alternative 12-Month Success
Description: Alternative 12-month success is defined as freedom from documented symptomatic AF/AT/AFL (of unknown origin) episodes based on electrocardiographic data (>=30 seconds on arrhythmia monitoring device) through the effectiveness evaluation period (Day 91 through Day 365) and freedom from the following failure modes: freedom from acute procedural failure, freedom from non-study catheter failure, freedom from repeat ablation failure, freedom from DC Cardioversion failure, freedom from recurrence (captured on 12-lead ECG) failure, and freedom from anti-arrhythmic drug failure. AFL of unknown origin is defined as all AFL except those CTI dependent AFL as confirmed by accepted EP maneuvers (e.g. entrainment or activation mapping) in an EP study.
Time Frame: From Day 91 up to Day 365 post-procedure (Day of procedure = Day 0)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 93 | 250
percentage of participants | 67.7 | 69.6

5. Secondary Outcome: Percentage of Participants With 12-Month Symptomatic Recurrence
Description: 12-month symptomatic recurrence endpoint is defined as freedom from documented symptomatic AF/AT/AFL (of unknown origin) episodes based on electrocardiographic data (>=30 seconds on arrhythmia monitoring device) through the effectiveness evaluation period (Day 91 through Day 365) in participants regardless of antiarrhythmic drug (AAD) use and freedom from the following failure modes: freedom from acute procedural failure, freedom from non-study catheter failure, freedom from repeat ablation failure, freedom from DC Cardioversion failure, and freedom from recurrence (captured on 12-lead ECG) failure. AFL of unknown origin is defined as all AFL except those CTI dependent AFL as confirmed by accepted EP maneuvers (e.g. entrainment or activation mapping) in an EP study.
Time Frame: From Day 91 up to Day 365 post-procedure (Day of procedure = Day 0)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 93 | 249
percentage of participants | 75.3 | 74.3

6. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Atrial Fibrillation Effect on Quality-of-Life (AFEQT) Scale Score
Description: AFEQT questionnaire is an atrial fibrillation-specific health-related quality of life (HRQoL) questionnaire designed to assess the impact of atrial fibrillation on participant's HRQoL. The questionnaire includes 20 questions on a 7-point Likert scale. Questions 1 to 18 evaluated HRQoL and questions 19 to 20 related to participant's satisfaction with treatment. Overall scores ranged from 0 to 100, where 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered). Therefore, a positive change in score corresponds to improvement in QoL. Total score was calculated using AFEQT formula: 100 minus ([sum of severity for all questions answered minus number of questions answered]*100 / total number questions answered*6).
Time Frame: Baseline, Month 12
Population: Roll-in arm: Roll-in analysis set defined as all participants who were enrolled in the roll-in phase and had undergone the RF delivery with the study catheters. Main study arm: mITT analysis set defined as enrolled participants who met eligibility criteria and had insertion of the Biosense Webster HELIOSTAR catheter. Here, 'N' (number of participants analyzed): participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 94 | 237
score on a scale | 33.37 (23.275) | 35.90 (21.754)

7. Secondary Outcome: Percentage of Participants With 12-Month Single Procedure Success
Description: 12-month single procedure success is defined as freedom from documented symptomatic AF/AT/AFL (of unknown origin) episodes based on electrocardiographic data (>=30 seconds on arrhythmia monitoring device) through the effectiveness evaluation period (Day 91 through Day 365) and freedom from the following failure modes: freedom from acute procedural failure, freedom from non-study catheter failure, freedom from repeat ablation failure, freedom from DC Cardioversion failure, freedom from recurrence (captured on 12-lead ECG) failure, and freedom from anti-arrhythmic drug failure. AFL of unknown origin is defined as all AFL except those CTI dependent AFL as confirmed by accepted EP maneuvers (e.g. entrainment or activation mapping) in an EP study.
Time Frame: From Day 91 up to Day 365 post-procedure (Day of procedure = Day 0)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Roll-in Phase | Main Study
Number analyzed (Participants) | 93 | 250
percentage of participants | 67.7 | 68.4

ADVERSE EVENTS:
Time Frame: From pre-procedure on Day 0 up to Month 12
Description: All-cause mortality: All enrolled roll-in phase participants and all-enrolled main study participants. Serious/other AEs: For main study, safety analysis set (enrolled participants who had insertion of study catheter); For roll-in phase, roll-in analysis set (all participants who were enrolled in the roll-in phase and had undergone the radiofrequency (RF) delivery with the study catheters).
Arm/Group | Roll-in Phase | Main Study
All-Cause Mortality (participants affected / at risk) | 0/117 | 2/280
Serious Adverse Events (participants affected / at risk) | 19/94 | 50/260
Other Adverse Events (participants affected / at risk) | 42/94 | 97/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roll-in Phase (N=94) | Main Study (N=260)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 11
Atrial flutter (Cardiac disorders) | 0 | 5
Atrial tachycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Contrast media reaction (Immune system disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Polymenorrhagia (Reproductive system and breast disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Iliac vein perforation (Vascular disorders) | 0 | 1
Internal haemorrhage (Vascular disorders) | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roll-in Phase (N=94) | Main Study (N=260)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 4
Atrial flutter (Cardiac disorders) | 5 | 8
Atrial tachycardia (Cardiac disorders) | 0 | 3
Atrioventricular block first degree (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 3
Pericarditis (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 2
Sinus arrest (Cardiac disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 2
Visual impairment (Eye disorders) | 2 | 2
Vitreous floaters (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Chronic gastritis (Gastrointestinal disorders) | 1 | 2
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0
Gastric hypomotility (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 3
Chest pain (General disorders) | 4 | 12
Fatigue (General disorders) | 3 | 2
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 6
Vessel puncture site haemorrhage (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 5
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Chemical burn (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 2
Oesophageal injury (Injury, poisoning and procedural complications) | 0 | 2
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 4
Chest X-ray abnormal (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 2
Heart sounds abnormal (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Computerised tomogram liver (Investigations) | 1 | 0
Haematocrit increased (Investigations) | 1 | 0
Haemoglobin increased (Investigations) | 1 | 0
Helicobacter test positive (Investigations) | 1 | 0
Laboratory test abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 2
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 2
Poor quality sleep (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 4
Haematuria (Renal and urinary disorders) | 1 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Blood pressure inadequately controlled (Vascular disorders) | 0 | 2
Essential hypertension (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 5
Hypertension (Vascular disorders) | 2 | 5
Hypotension (Vascular disorders) | 1 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning the study, investigational medical device, sponsor operations, patent application, manufacturing processes, and basic scientific data supplied by the sponsor to the investigator and not previously published, are considered confidential and remain the sole property of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03683030/Prot_004.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03683030/SAP_005.pdf